CLINICAL TRIAL: NCT03243175
Title: Avoiding Anticoagulation After IntraCerebral Haemorrhage
Acronym: A3ICH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016_77; 2017-004371-31 (EudraCT Number)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Intracerebral Hemorrhage; Atrial Fibrillation; Microhaemorrhage
Keywords: intracerebral hemorrhage; atrial fibrillation; microhemorrhage; oral anticoagulation; left atrial appendage closure
MeSH Terms: conditions — Cerebral Hemorrhage; Atrial Fibrillation | interventions — apixaban; Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: 1:1:1
Who Masked: Outcomes Assessor
Masking Description: PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Direct Oral Anticoagulant (DOAC) (Experimental): Apixaban 5MG twice daily
  Interventions: Drug: Apixaban 5 MG
- Left Atrial Appendage Closure (LAAC) (Experimental): Devices will be chosen by local teams.
  Interventions: Device: left atrial appendage closure
- Control (No Intervention): avoiding anticoagulation and LAAC during the entire study period The standard clinical practice without OAC may include: antiplatelet drug (in case of comorbidities such as coronary heart disease) or no antithrombotic drug

INTERVENTIONS:
Drug: Apixaban 5 MG — Apixaban 5mg x 2 during 24 months
  Other Names: ELIQUIS 5mg
  Arms: Direct Oral Anticoagulant (DOAC)
Device: left atrial appendage closure — left atrial appendage closure
  Arms: Left Atrial Appendage Closure (LAAC)

SUMMARY:
Randomised controlled trials (RCTs) demonstrate a substantial benefit from oral anticoagulant drugs for the prevention of stroke and systemic embolism in non-valvular atrial fibrillation (AF). However, these RCTs excluded patients with prior intracerebral haemorrhage (ICH). Therefore, guidelines are unable to recommend whether oral anticoagulant drugs, in particular non-vitamin K antagonist (called direct OAC) - can be used for patients with AF after an intracerebral haemorrhage.

Roughly 30% of adults with ICH have AF but in 2017 it remains unclear whether they should start oral anticoagulant drugs, be treated with left atrial appendage closure (LAAC) or avoid anticoagulation and LAAC.

DETAILED DESCRIPTION:
Open label randomised controlled multicentre clinical trial with masked outcome assessment (PROBE design) comparing 3 strategies (1:1:1): anticoagulation with a Direct OAC (Apixaban 5mgx2/day) vs avoid anticoagulation with left atrial appendage closure (LAAC) compared to usual care (avoid anticoagulation).

Primary outcome: the net clinical benefit (composite outcome of major ischaemic and haemorrhagic events) during a follow-up of 24 months (adjudication committee masked to the randomisation arm

The results of A3ICH will help the clinician to decide which strategy is the most effective in terms of benefit/risk ratio to prevent the risk of stroke or systemic embolism in patients with a history of ICH and AF. A3ICH will address this increasingly common dilemma and could affect clinical practice.

Data from A3ICH will contribute to an international individual patient data meta-analysis.

ELIGIBILITY:
Inclusion criteria

* Adult (older than 18 years old, no upper age limit)
* with a history of paroxysmal, persistent or long-standing non-valvular atrial fibrillation (documented on an electrocardiogram)
* and a CHA2DS2VASc score of 2 or more who have an indication for long-term anticoagulation
* who suffered from a spontaneous intracerebral haemorrhage (while being treated with oral anticoagulants or not) documented with brain CT or MRI
* more than 14 days before randomization (no upper delay limit)
* for whom there is a clinical equipoise regarding the choice of the best preventive strategy to avoid future vascular events.

Exclusion criteria for all treatment groups

* Pre-randomisation modified Rankin score of 4 or 5
* Conditions other than atrial fibrillation for which the patient requires long term anticoagulation (for example prosthetic mechanical heart valve)
* Serious bleeding events within the 6 months before randomisation (except for intracerebral haemorrhage)
* Life expectancy of less than 1 year
* Pregnancy or breastfeeding

Exclusion criteria related to the LAAC only

* Contraindications due to local, anatomical reasons (such as thrombus in the left atrial appendage, infection with a risk of endocarditis)
* Patients older than 85 years
* CHA2DS2VASc score of 2 or 3
* Patient or attending physician are unwilling to undergo/perform intervention for LAAC

Exclusion criteria related to the Direct OAC only

* Chronic renal insufficiency (clearance of creatinine by Cockcroft method < 30ml/min)
* Body weight lower than 50 kg
* Allergy to apixaban
* Coexisting conditions predisposing to head trauma (e.g. gait disturbances, uncontrolled seizures disorders)
* Patient or attending physician are unwilling to use of Direct OAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Composite of all fatal or non-fatal major cardiovascular/cerebrovascular ischaemic or haemorrhagic intracranial/extracranial events | within 24 months after randomization.
  The composite endpoint will enable to evaluate the net clinical benefit of the different therapeutic strategies.
  Definition of fatal event: when death is occurring within 30 days after the events.

SECONDARY OUTCOMES:
Each individual component of the composite outcome (fatal or non-fatal major cardiovascular/cerebrovascular ischaemic or haemorrhagic intracranial/extracranial events). | at 12 and 24 months after randomization
  fatal or non-fatal major cardiovascular/cerebrovascular ischaemic or haemorrhagic intracranial/extracranial events).
Death of any cause | at 12 and 24 months after randomization
  death
Modified Rankin Scale | at 12 and 24 months after randomization
  functional dependence
EQ-5D (EuroQoL) Score | at 12 and 24 months after randomization
  health-related quality of life
neuroradiological biomarkers | Baseline
  on brain MRI
Complications of endovascular treatment | up to 30 days
  including device related complications

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Cordonnier, MD, PhD, Principal Investigator — University Hospital Lille, Inserm, Univ Lille
Locations (3):
- France (3):
  - Hôpital Roger Salengro, CHU, Lille
  - GHICL, Lomme
  - CH De Tourcoing, Tourcoing

IPD SHARING:
Plan to Share IPD: Yes
Prof Cordonnier (chief investigator of A3ICH) is a member of the international Collaboration Of Controlled Randomised trials of Oral Antithrombotic drugs after intraCranial Haemorrhage (COCROACH - coordination Prof Rustam Al-Shahi Salman, UK) working towards a pre-planned individual patient data meta-analysis
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170